CLINICAL TRIAL: NCT07094659
Title: Aging and Task-Specific Training to Reduce Falls
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0959; 2R01AG050672-06A1 (NIH)
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Fall Prevention
Keywords: balance; fall risk; fall prevention; slips; trips; older adults; reactive balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Task-Specific Balance Training (Experimental): Participants in the task-specific balance training group will receive 8 weeks of task-specific balance training that includes both functional tasks and predictable perturbations specific to slips and trips. Sessions will be completed 2x per week for 8 weeks (16 sessions total).
  Interventions: Behavioral: Task-Specific Balance Training
- Treadmill Perturbation Training (Active Comparator): Participants in the treadmill perturbation training group will receive 8 weeks of training that includes exposure to slip-like and trip-like perturbations delivered via motorized treadmill. Sessions will be completed 2x per week for 8 weeks (16 sessions total).
  Interventions: Behavioral: Treadmill Perturbation Training
- Conventional Balance Training (Active Comparator): Participants in the conventional balance training group will receive 8 weeks of training that includes conventional exercises designed to improve balance control. Sessions will be completed 2x per week for 8 weeks (16 sessions total).
  Interventions: Behavioral: Conventional Balance Training

INTERVENTIONS:
Behavioral: Task-Specific Balance Training — Participants in the intervention groups will receive 8 weeks of task-specific balance training that includes both functional tasks and predictable perturbations specific to slips and trips. Sessions will be completed 2x per week for 8 weeks (16 sessions total).
  Arms: Task-Specific Balance Training
Behavioral: Treadmill Perturbation Training — Participants in the treadmill perturbation training group will receive 8 weeks of training that includes exposure to slip-like and trip-like perturbations delivered via motorized treadmill. Sessions will be completed 2x per week for 8 weeks (16 sessions total).
  Arms: Treadmill Perturbation Training
Behavioral: Conventional Balance Training — Participants in the conventional balance training group will receive 8 weeks of training that includes conventional exercises designed to improve balance control. Sessions will be completed 2x per week for 8 weeks (16 sessions total).
  Arms: Conventional Balance Training

SUMMARY:
The goal of this clinical trial is to examine the effects of a novel task-specific balance training for reducing environmental falls in community ambulatory older adults who are at-risk of falling. The main questions it aims to answer are:

* Does task-specific balance training improve the ability to prevent falling when unexpected perturbations such as slips and trips occur, and/or improve balance control during self-initiated movements?
* Does task-specific balance training reduce real-life falls for 18 months after training?

Researchers will compare task-specific balance training with conventional balance training and treadmill perturbation-based training to examine how this novel intervention compares to established interventions for improving balance.

Participants who participate in the study will be asked to do the following:

* Complete a pre-training assessment of their balance control, and then be randomized to one of three training groups: 1) task-specific balance training, 2) treadmill perturbation-based training, and 3) conventional balance training
* Complete their assigned training protocol for 8 weeks (2x per week for a total of 16 sessions)
* Complete 2 post-training assessments of their balance control, the first being completed immediately after the training is completed, and the second being completed 18 months after the training is completed
* Wear a physical activity monitor for 18 months after completing the intervention to monitor their real life falls.

DETAILED DESCRIPTION:
The proposed study employs a randomized, controlled design to assess the immediate and long-term effects of task-specific balance training for reducing environmental falls in at-risk community-ambulatory older adults. >33% of older adults fall at least once each year, leading to serious injuries (e.g., hip fractures), comorbidities (e.g., Alzheimer's Disease and related dementias), and higher chances of falling again. Most falls occur due to environmental disturbances which cause a loss of balance while walking (i.e., slips, trips). Our lab has established that overground perturbation training (repeated exposure to unpredicted perturbations) improves balance control in both predictable (i.e., volitional/anticipatory) and unpredictable (i.e., reactive) environments, and reduces real-life falls among older adults. However, overground perturbation training is not suitable for routine clinical application due to its complex design, space, and technology requirements. An alternative method for delivering perturbation training is via commercial treadmill systems, which enhance fall-resisting skills and are more feasible for community-translation. However, treadmill perturbation training still requires costly equipment and has lower translational effectiveness for reducing falls in community-ambulatory older adults than overground training. This may be because treadmill perturbation training mainly trains reactive balance control, while falls may also occur due to deficits in volitional balance control which affect gait stability during daily tasks. Volitional balance training has primarily comprised of conventional balance exercises delivered as a part of physical rehabilitation; however, conventional balance exercises generally do not translate to improvements in reactive balance control when exposed to unpredicted perturbations and have limited effects on reducing real-life falls. A fall prevention intervention that targets both volitional and reactive balance control could more effectively reduce falls in at-risk older adults than existing paradigms which only train a single domain (e.g., reactive-dominant treadmill perturbation training or volitional-dominant conventional balance training). We have developed a novel balance training program that includes both volitional-based task-specific exercises and reactive-based predictable perturbations to target the strategies involved in preventing slip- and trip-falls. This task-specific balance training requires little set-up and equipment, making it cost-effective, feasible and accessible. We will examine the immediate effects of 8 weeks (16 sessions) of task-specific balance training on reactive balance (Aim 1) and volitional balance (Aim 2), compared with established fall prevention paradigms (treadmill perturbation training and conventional balance training). Additionally, we will evaluate the longer-term retention (18 months) of task-specific balance training and effects on real-life falls and falls efficacy (Aim 3). In an exploratory aim, we will also examine the neuromuscular adaptations induced through training using muscle synergy analysis (Aim 4). If successful, our novel intervention could be implemented as a feasible, safe, and effective fall prevention intervention, with large potential for direct dissemination to clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 90 years of age to include community dwelling older adults
* Understand English to ensure ability to safely complete study protocols
* Able to walk independently for 1 block and 10 meters without an assistive device to ensure ability to complete exercises and reactive balance assessments
* 'At-risk' adults: Participants who report experience of at least 1 fall in the past 12 months or participants who are categorized as at high fall- risk using our fall risk prediction model which can predict the risk of both slip and trip related falls.

Exclusion Criteria:

* Major surgery less than 6 months ago to avoid complications due to training
* Hospitalization less than 3 months ago to avoid complications due to training
* Taking any sedative drugs to avoid interference with training
* Acute or uncontrolled neurological or cardiopulmonary or musculoskeletal or cancer diagnosis to avoid complications due to training
* Have intact visual and auditory ability with or without corrective aids to avoid confounding effects on balance
* Severe osteoporosis measured by a score of less than negative two point five on heel bone density scan to avoid complications due to training
* Loss of sensation on monofilament test to avoid confounding effects on outcome assessments
* Cognitive impairment indicated by a score of less than 25 out of 30 on the mini mental state exam to ensure ability to follow instructions for safety
* Shortness of breath or uncontrolled pain higher than a three out of ten or inability to achieve age specified minimal distance on the 6 minute walk test for endurance to avoid complications due to training

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Reactive Stability | Immediately post and at 18 months
  Center of mass position will be computed via Helen Hayes marker set using an eight-camera motion capture system and normalized by foot length. The center of mass velocity will be computed by the first order derivative of the center of mass position and normalized to acceleration due to gravity and participant's body height. Reactive stability will be calculated as the shortest perpendicular distance from the center of mass state (position and velocity) to the dynamic feasible theoretical boundary for loss of balance. Reactive stability values less than 0 indicate greater instability in the backward direction, while values greater than 1 indicate greater instability in the forward direction.
Vertical Limb support | Immediately post and at 18 months
  Limb support will be quantified by change in vertical limb support upon the perturbation hip height. The hip height, Zhip, will be obtained as the vertical distance of the bilateral hip midpoint to the surface of the platform. Its positive direction is upward. Zhip will be normalized to bh. Change in Zhip at recovery foot touchdown and its minimum value post-perturbation from its pre-perturbation value will be extracted.
Laboratory falls | Immediately post and at 18 months
  Falls on laboratory perturbation will be identified when the peak load cell force, which is attached to the full-body safety harness exceeds 30% of participant body weight. This will further be verified by video recordings.
Functional Gait Assessment | Baseline, Immediately post and at 18 months
  The functional gait assessment assesses dynamic postural stability and the ability to perform multiple motor tasks during walking, including 10 items where the researcher rates the participant's ability (from 0-3) to perform 10 different gait tasks, such as walking with the eyes closed, walking up stairs, and walking with changes in gait speed. We selected the FGA to determine training-induced improvements in volitional balance control as it highly mimics scenarios which might be encountered during ambulation in daily living.
Real-life falls | Recorded retrospectively (12 months before training) and weekly for 18 months post-training
  Participants will be sent a weekly text inquiring if they experienced a fall or loss of balance that day. If participants respond "yes," they will be followed up with a phone call to inquire about fall details. Participants can also choose to mail in fall logs if they opt out of weekly messaging. Real-life fall data will also be supplemented with daily device-recording using wrist-worn ActiGraph Accelerometers.
Activities-specific Balance Confidence Scale (ABC) | Baseline, Immediately post and at 18 months
  Falls efficacy will be assessed using the Activities-Specific Balance Confidence Scale (ABC), which asks individuals to rate their level of confidence (0-100%) that they will not lose their balance while performing various activities of daily living, such as getting onto an escalator or reaching into a cabinet. An overall score of 0% indicates no confidence, while a score of 100% indicates complete confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT07094659/Prot_SAP_000.pdf